CLINICAL TRIAL: NCT02855151
Title: EUS for Gastrointestinal Disorders: a Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1497
Record Dates: First submitted 2016-07-18; First posted 2016-08-04 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: GI Tract Disorders; Pancreatic Disorders; EUS
Keywords: EUS
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the EUS registry is to record information about Endoscopic Ultrasound (EUS) on the management of gastrointestinal disease. The registry will evaluate efficacy, safety and technical success of the Endoscopic Ultrasound (EUS). Design is retrospective and prospective registry study.

ELIGIBILITY:
Inclusion Criteria:

* All patients submitted to EUS,
* Informed consent.

Exclusion Criteria:

* Age less than 18 y
* Patient who did not give the consent to the processing of personal data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients submitted to diagnostic or therapeutic EUS
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-01; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | 2 days
  Documentation of adverse events.

SECONDARY OUTCOMES:
Diagnostic yied of elastography during EUS | 0 Day
  sensitivity and specificity of EUS with elastography
Diagnostic yied of Contrast-Enhanced Endoscopic Ultrasonography | 0 Day
  sensitivity and specificity contrast medium
Tissue acquisition during EUS | 0 Days
  sensitivity and specificity of tissue acquisition

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — Humanitas University; Silvia Carrara, MD, Study Director — Humanitas Cancer Center
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carrara S, Rahal D, Khalaf K, Rizkala T, Koleth G, Bonifacio C, Andreozzi M, Mangiavillano B, Auriemma F, Bossi P, Balzarotti M, Facciorusso A, Staiano T, Maldi E, Spadaccini M, Colombo M, Fugazza A, Maselli R, Hassan C, Repici A. Diagnostic accuracy and safety of EUS-guided end-cutting fine-needle biopsy needles for tissue sampling of abdominal and mediastinal lymphadenopathies: a prospective multicenter series. Gastrointest Endosc. 2023 Aug;98(2):191-198. doi: 10.1016/j.gie.2023.03.018. Epub 2023 Mar 27. PMID 36990125
- [Derived] Carrara S, Di Leo M, Grizzi F, Correale L, Rahal D, Anderloni A, Auriemma F, Fugazza A, Preatoni P, Maselli R, Hassan C, Finati E, Mangiavillano B, Repici A. EUS elastography (strain ratio) and fractal-based quantitative analysis for the diagnosis of solid pancreatic lesions. Gastrointest Endosc. 2018 Jun;87(6):1464-1473. doi: 10.1016/j.gie.2017.12.031. Epub 2018 Jan 9. PMID 29329992